CLINICAL TRIAL: NCT02048332
Title: Donor-Derived Viral Specific T-cells (VSTs) for Treatment of Viral Infections After Allogeneic Stem Cell Transplant
Brief Title: Donor-Derived Viral Specific T-cells (VSTs)
Acronym: VSTs
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Hoxworth Blood Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-2777
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Allogeneic Stem Cell Transplant; Viral Infection; Viral Reactivation
Keywords: Epstein-Barr Virus (EBV); Adenovirus (ADV); t-cells; donor; transplant; children; cytomegalovirus (CMV); BK virus (BKV)
MeSH Terms: conditions — Virus Diseases; Epstein-Barr Virus Infections; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Viral Specific VST Infusion (Experimental): Viral reactivation or infection. VST Reinfusion required.
  Interventions: Biological: Viral specific VST Infusion

INTERVENTIONS:
Biological: Viral specific VST Infusion — VSTs will be infused into stem cell transplant recipients who have evidence of viral infection or reactivation defined as any of the below:
  * Blood adenovirus PCR ≥ 1,000
  * Blood CMV PCR ≥ 500
  * Blood EBV PCR ≥ 9,000
  * Plasma BKV PCR >1,000
  * Plasma JC Virus PCR >1,000
  * Evidence of invasive adenovirus infection or disease, defined as the presence of adenoviral positivity in one or more sites.
  * Evidence of invasive CMV infection, eg pneumonitis, retinitis, colitis
  * Evidence of invasive EBV disease/infection, EBV-associated lymphoproliferation (EBV-LPD) defined as proven EBV-LPD by biopsy or probable EBV-LPD defined as an elevated EBV DNA level in the blood associated with clinical symptoms (adenopathy or fever or masses on imaging) but without biopsy confirmation, or EBV-associated malignancies.
  * Evidence of symptomatic BK virus infection, which may include symptomatic hemorrhagic cystitis, or BK nephropathy.
  * Evidence of PML or other CNS infection due to JC virus.

SUMMARY:
In this research study, the investigators want to learn more about the use of donor-derived viral specific T-cells (VSTs) to treat viral infections that occur after allogeneic stem cell transplant. A viral specific T cell is a T lymphocyte (a type of white blood cell) that kills cells that are infected (particularly with viruses). Allogeneic means the stem cells come from another person. These VSTs are cells specially designed to fight the virus infections that can happen after a bone marrow transplant.

The investigators are asking people who have undergone or will undergo an allogeneic stem cell transplant to enroll in this research study, because viral infections are a common problem after allogeneic stem cell transplant and can cause significant complications including death.

Stem cell transplant reduces a person's ability to fight infections. There is an increased risk of getting new viral infections or reactivation of viral infections that the patient has had in the past, such as cytomegalovirus (CMV), Epstein-Barr virus (EBV), adenovirus (ADV), BK virus (BKV), and JC virus. There are anti-viral medicines available to treat these infections, though not all patients will respond to the standard treatments. Moreover, treatment of viral infections is expensive and time consuming, with families often administering prolonged treatments with intravenous anti-viral medications, or patients requiring prolonged admissions to the hospital. The medicines can also have side effects like damage to the kidneys or reduction in the blood counts, so in this study the investigators are trying to find an easier way to treat these infections.

DETAILED DESCRIPTION:
The stem cell matched donor will be asked to provide a blood donation for the VSTs generation. In the laboratory, the investigators will treat this blood sample to select out the cells that will help fight viruses. The cells will be grown with peptides (protein fragments that represent parts of the virus that will encourage the donor immune cells to grow). The cells will be grown in the laboratory so that there is a stock of virus fighting cells for the patient to use in the future. The investigators will freeze the cells and store them in a freezer in the laboratory.

If the patient has signs of virus in their blood after the transplant, they will be given the cells to help fight the infection. If there are signs that the cells are helping fight the infection, more cells may be given. The patient may get the cells up to 5 times, with 21 days between each treatment (this timeframe may be shortened to 14 days for patients with no evidence of viral response). If the patient does not show signs of a virus, the cells will stay in the freezer.

Following VST infusion, (s)he will be monitored with physical exams daily while inpatient and weekly while outpatient as well as blood tests weekly until 30 days after the last infusion of cells. The patient will have 3 teaspoons (15 mL) of blood drawn and urine collected before each cell infusion and then once a week after each infusion for 4 weeks and then once a month if possible for 1 year after the last infusion, all to monitor for the viral response.

ELIGIBILITY:
Inclusion Criteria:

* Recipient must be at least 21 days after stem cell infusion
* Clinical status must allow tapering of steroids to 0.5mg/kg prednisone or other steroid equivalent
* Recipient must have achieved engraftment with ANC ≥ 500

Exclusion Criteria:

* Active acute GVHD grades II-IV
* Uncontrolled bacterial or fungal infection
* Uncontrolled relapse of malignancy requiring treatment with chemotherapy
* Infusion of ATG or alemtuzumab within 2 weeks of VST infusion

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2014-02-05 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Successful production of viral specific T-cells | Within 30 days post culture initiation
  Of the patients who had a VST culture initiated, successful production of VST cells is defined as meeting the protocol-defined release criteria.
Percentage of patients who do not have infusional toxicity | Through 30 minutes post infusion
  Patients will be monitored for infusional toxicity
Incidence of GVHD associated with VST infusion | Through 30 days after infusion
  Patients will be monitored for the development of VST associated GVHD

SECONDARY OUTCOMES:
Presence of viral-specific T-cells | At 30 days after infusion
  Presence of viral-specific T-cells in the participant's blood will be assessed by Elispot assay
Viral burden | At 30 days after infusion
  The viral burden will be assessed using the protocol-defined efficacy assessment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Grimley, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - Akron Children's Hospital, Akron, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

REFERENCES:
- [Derived] Galletta TJ, Lane A, Lutzko C, Leemhuis T, Cancelas JA, Khoury R, Wang YM, Hanley PJ, Keller MD, Bollard CM, Davies SM, Grimley MS, Rubinstein JD. Third-Party and Patient-Specific Donor-Derived Virus-Specific T Cells Demonstrate Similar Efficacy and Safety for Management of Viral Infections after Hematopoietic Stem Cell Transplantation in Children and Young Adults. Transplant Cell Ther. 2023 May;29(5):305-310. doi: 10.1016/j.jtct.2023.01.027. Epub 2023 Feb 3. PMID 36736781
- [Derived] Rubinstein JD, Zhu X, Leemhuis T, Pham G, Ray L, Emberesh S, Jodele S, Thomas S, Cancelas JA, Bollard CM, Hanley PJ, Keller MD, Grimley O, Clark D, Clark T, Lindestam Arlehamn CS, Sette A, Davies SM, Nelson AS, Grimley MS, Lutzko C. Virus-specific T cells for adenovirus infection after stem cell transplantation are highly effective and class II HLA restricted. Blood Adv. 2021 Sep 14;5(17):3309-3321. doi: 10.1182/bloodadvances.2021004456. PMID 34473237